CLINICAL TRIAL: NCT01978782
Title: Pharmacokinetic Drug-drug Interaction Study Between RaltEgravir and CITALopram in Healthy Subjects (RECITAL).
Acronym: RECITAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF12.04; 2012-005148-50 (EudraCT Number)
Record Dates: First submitted 2013-10-22; First posted 2013-11-08 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2015-07

CONDITIONS: HIV; Depression
Keywords: raltegravir; citalopram; pharmacokinetics; drug-drug interaction
MeSH Terms: conditions — Depression | interventions — Raltegravir Potassium; Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- raltegravir alone (Active Comparator): raltegravir 400 mg BID for 5 days
  Interventions: Drug: raltegravir
- citalopram alone (Active Comparator): citalopram 10 mg QD for 3 days, followed by citalopram 20 mg QD for 13-14 days
  Interventions: Drug: citalopram
- raltegravir + citalopram (Experimental): raltegravir 500 mg BID and citalopram 20 mg QD for 5 days
  Interventions: Drug: raltegravir; Drug: citalopram

INTERVENTIONS:
Drug: raltegravir
  Other Names: isentress
  Arms: raltegravir + citalopram; raltegravir alone
Drug: citalopram
  Arms: citalopram alone; raltegravir + citalopram

SUMMARY:
Depression is the most common mental health disorder among HIV-patients. Recognizing and treating depression is important in order to improve quality of life and health outcomes in those living with HIV. In clinical practice selective serotonin reuptake inhibitors (SSRIs) are used most frequently in HIV patients with depressive symptoms. A complicating factor in the concomitant use of antiretroviral agents and antidepressant therapy is the occurrence of drug-drug interactions. Citalopram can be seen as one of the preferred SSRIs in HIV-infected patients because citalopram has a relatively favourable drug interaction profile compared to other SSRIs. Raltegravir is an HIV-1 integrase inhibitor and is frequently being used as antiretroviral agent in combination with tenofovir/emtricitabine in HIV-patients. Raltegravir has shown sustained antiretroviral activity, is generally well tolerated and has little propensity to interact with other drugs because it does not inhibit or induce CYP450 enzymes. Theoretically, no clinically relevant drug interaction is expected between raltegravir and citalopram as raltegravir is not a CYP2D6 substrate and thus will not be affected by the possible inhibition of CYP2D6 by citalopram. Raltegravir is metabolized by UGT but citalopram is not known to influence UGT. A possible interaction may occur through inhibition of P-gp mediated transport of raltegravir by citalopram. However, even when no drug interaction is expected theoretically, it may be recommended to collect sufficient clinical evidence to support this hypothesis because unexpected interactions with raltegravir have been observed in the past. In order to be able to recommend raltegravir and citalopram concomitant use, a pharmacokinetic study in healthy volunteers is proposed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 and not older than 55 years at screening.
2. Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to Day 1.
3. Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
4. Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
5. Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry, haematology and urinalysis testing within 4 weeks prior to Day 1. Results of biochemistry, haematology and urinalysis testing should be within the laboratory's reference ranges. If laboratory results are not within the reference ranges, the subject is included on condition that the Investigator judges that the deviations are not clinically relevant. This should be clearly recorded.
6. Subject has a normal blood pressure and pulse rate, according to the Investigator's judgement.

Exclusion Criteria:

1. Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
2. Positive HIV test.
3. Positive hepatitis B or C test.
4. Pregnant female (as confirmed by an hCG test performed less than 4 weeks before day 1) or breast-feeding female. Female subjects of childbearing potential without adequate contraception, e.g. hysterectomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout the entire conduct of the study.
5. Therapy with any drug (for two weeks preceding Day 1), except for acetaminophen.
6. Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disorders, renal and hepatic disorders, hormonal disorders (especially diabetes mellitus), coagulation disorders.
7. Relevant history or presence of QT syndrome, prolonged QTc time, bradycardia, hypokalaemia or hypomagnesaemia, recent acute myocardial infarction, or uncompensated heart failure.
8. Relevant history or current condition that might interfere with drug ab-sorption, distribution, metabolism or excretion.
9. History of or current abuse of drugs, alcohol or solvents.
10. Inability to understand the nature and extent of the study and the pro-cedures required.
11. Participation in a drug study within 60 days prior to Day 1.
12. Donation of blood within 60 days prior to Day 1.
13. Febrile illness within 3 days before Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
raltegravir AUC and citalopram AUC | at steady state: day 5 of raltegravir treatment and day 16 or later for citalopram
  To assess the effect of multiple dose citalopram on the steady state pharmacokinetics of raltegravir and vice versa by intrasubject comparison in healthy subjects.
  * The comparison of steady state raltegravir (400 mg BID for 5 days) pharmacokinetics (AUC0-12h, Cmax, C12h) with steady state citalopram (20 mg QD) vs. raltegravir alone by intrasubject comparison.
  * The comparison of steady state citalopram (20 mg QD) pharmacokinetics (AUC0-24h, Cmax, C24h) with steady state raltegravir (400 mg BID) vs. citalopram alone by intrasubject comparison.

SECONDARY OUTCOMES:
Adverse Events | up to approximately 13 weeks (from screening until the last study visit)
  Adverse events will be scored and laboratory measurements for safety will be collected frequently from screening onwards (maximum 4 weeks before the start of the study) until the last study visit (Day 60) or longer if applicable.

CONTACTS AND LOCATIONS:
Locations (1):
- CRCN Radboud university medical center, Nijmegen, Netherlands

REFERENCES:
- [Result] Blonk MI, Langemeijer CC, Colbers AP, Hoogtanders KE, van Schaik RH, Schouwenberg BJ, Burger DM. Pharmacokinetic drug-drug interaction study between raltegravir and citalopram. Antivir Ther. 2016;21(2):143-52. doi: 10.3851/IMP2993. Epub 2015 Sep 16. PMID 26375942
- See also: Abstract 53: Pharmacokinetic drug-drug interaction study between raltegravir and citalopram in healthy volunteers. — http://regist2.virology-education.com/abstractbook/2015_4.pdf
- See also: paper — https://pubmed.ncbi.nlm.nih.gov/26375942/